CLINICAL TRIAL: NCT06851156
Title: An Exploratory Trial Evaluating Temporal Interference Stimulation of CM-pf In Patients With Disorders of Consciousness
Brief Title: Transcranial Temporal Interference Stimulation In Severely Brain Injured Patients With Disorders of Consciousness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20242231jiangwen
Record Dates: First submitted 2025-02-18; First posted 2025-02-28 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-02

CONDITIONS: Disorders of Consciousness; Severe Brain Injury; Unresponsive Wakefulness Syndrome; Minimally Conscious State
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries; Persistent Vegetative State

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transcranial Temporal Interference Stimulation (Experimental): tTIS is applied over the bilateral CM-pf for 10 days, once a day.
  Interventions: Device: tTIS

INTERVENTIONS:
Device: tTIS — CM-pf tTIS

SUMMARY:
The purpose of this academic lead study is to explore the effect of noninvasive neuromodulation of the CM-pf via tTIS for patients with disorders of consciousness.

ELIGIBILITY:
Inclusion Criteria:

* traumatic and nontraumatic etiology of VS/UWS or MCS according to published diagnostic criteria.

Exclusion Criteria:

* patients in coma, with less than 1 week after acute brain insult, with fluctuating diagnosis on baseline assessment, and with a metallic cerebral implant or pacemaker, and with epilepsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
CRS-R total score changes | From enrollment to the end of treatment at 10 days
  Coma Recovery Scale-Revised scale score, with score ranging from 0 to 23, was used to evaluate the consciousness condition.

SECONDARY OUTCOMES:
Numbers of patients with improved consciousness | From enrollment to the end of treatment at 10 days
EEG changes | From enrollment to the end of treatment at 10 days
  EEG power spectra, Connectivity and ABCD model, etc

CONTACTS AND LOCATIONS:
Overall Officials: wen Jiang, phD, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided